CLINICAL TRIAL: NCT01263145
Title: Phase Ib Dose Escalation and Biomarker Study of MK-2206 in Combination With Standard Doses of Weekly Paclitaxel in Patients With Locally Advanced or Metastatic Solid Tumors With an Expansion in Advanced Breast Cancer
Brief Title: MK2206 and Paclitaxel in Treating Patients With Locally Advanced or Metastatic Solid Tumors or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02562; NCI-2011-02562 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0245; CDR0000690723; 2010-0245 (Other: M D Anderson Cancer Center); 8739 (Other: CTEP); P30CA016672 (NIH); U01CA062461 (NIH); U01CA062490 (NIH)
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Adult Solid Neoplasm; Recurrent Breast Carcinoma; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — MK 2206; Paclitaxel

ARMS (1):
- Treatment (Akt inhibitor MK2206 and paclitaxel) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and Akt inhibitor MK2206 PO QD on days 2, 9, and 16. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of Akt inhibitor MK2206 (MK2206) when given together with paclitaxel and to see how well they work in treating patients with solid tumors that have spread to other places in the body and usually cannot be cured or controlled with treatment or breast cancer that has spread to other places in the body. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving Akt inhibitor MK2206 and paclitaxel may be a better treatment for solid tumors or breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of the combination of MK-2206 and weekly paclitaxel. (Dose-escalation phase) II. To determine the safety and anti-tumor activity of the combination in metastatic breast cancer. (Expansion phase)

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics of MK-2206 and weekly paclitaxel used in combination.

II. To determine the safety of MK-2206 and weekly paclitaxel used in combination.

III. To evaluate the toxicities and tolerability of the combination. IV. To document anti-tumor activity. V. To determine baseline molecular markers that may predict clinical activity. VI. To determine pharmacodynamic markers in blood and tumor tissue that may predict an increase in apoptosis (by cleaved caspase 3) and clinical activity.

VII. To determine concordance of phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) and phosphatase and tensin homolog (PTEN) status between primary tumor and distant metastasis.

VIII. To determine concordance of PIK3CA status of circulating tumor cells and distant metastasis.

OUTLINE: This is a dose-escalation study of Akt inhibitor MK2206.

Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15 and Akt inhibitor MK2206 orally (PO) once daily (QD) on days 2, 9, and 16. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors who have received at least two lines of therapy; for the expansion phase: female patients with metastatic breast cancer who have received a maximum of three lines of therapy
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelets >= 100,000/uL
* Hemoglobin (Hgb) >= 9 g/dL
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Prothrombin time (PT) within institutional guideline for biopsy procedure
* Total bilirubin =< 1.5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN (=< 3 x ULN for subjects with liver involvement with cancer)
* A known diabetic patient who is taking insulin or oral anti-diabetic therapy must have a hemoglobin A1C (HBA1C) =< 8% or a fasting serum glucose =< 110% ULN
* Patient will have a tumor suitable for fine-needle aspirates (FNA) and core biopsy for research purposes (determined by the treating physician)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) or evaluable disease (e.g., bone metastasis or lesions which do not fulfill RECIST criteria for metastatic disease)
* Patients with central nervous system (CNS) metastasis who have completed a course of therapy (for treatment of CNS metastasis) would be eligible for the study provided they are clinically stable for 1 month prior to entry as defined as:

  * No evidence of new or enlarging CNS metastasis
  * Off steroids and anticonvulsants
* Corrected QT (QTc) interval =< 450 msec (Bazett's formula)
* Negative serum pregnancy test beta-human chorionic gonadotropin (hCG) for patients of childbearing age
* For the dose escalation cohorts, patients must have received front-line, cytotoxic, systemic therapy (combination or single agent, with or without the addition of targeted agents) for advanced cancer
* For the expansion cohort, patients must have received no more than three lines of cytotoxic systemic therapy (combination or single agent, with or without the addition of targeted agents) for metastatic breast cancer; patients could have received paclitaxel in the adjuvant setting, but not in the metastatic setting
* The last line of therapy must have been administered > 21 days prior to initiation of treatment on this study
* Women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Both men and women and members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients taking a potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitor or inducer will be excluded; patients who have discontinued any of these medications must have a wash-out period of at least 5 days or at least 5 half-lives of the drug (whichever is longer) prior to the first dose MK-2206
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, bradycardia, related to cardiac disease, bundle branch block, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-01-05 (Actual); Primary Completion 2012-10-19 (Actual); Study Completion 2012-10-19 (Actual)

PRIMARY OUTCOMES:
Antitumor activity of the combination in metastatic breast cancer (Expansion phase) | Up to 3 weeks after completion of study treatment
MTD of the combination of MK-2206 and paclitaxel defined as the dose level in which less than or equal to 1 out of 6 patients develop dose limiting toxicity assessed using Common Terminology Criteria for Adverse Events version 4 (Phase I) | 21 days

SECONDARY OUTCOMES:
Change in average number of circulating tumor cells (CTCs) | Baseline to up to 2 weeks
  Will be determined by chi-square analysis or Fisher's Exact test and compared by Student t-test.
Change in multiplex proteomics | Baseline to up to day 17
Change in percentage of biomarkers assessed using immunohistochemistry | Baseline to up to 2 weeks
Change in percentage of marker of proliferation Ki-67 (Ki-67) positive cells | Baseline to up to 2 weeks
  Will be calculated using a two-sided one-sample t-test, at a significance level of 0.05.
Change in reverse phase proteomic arrays (RPPA) | Baseline to up to day 8
  Will be analyzed using the Wilcoxon rank test.
Pharmacokinetic parameters of Akt inhibitor MK2206 | On days 1-3, 5, 8, 16, 17, and 19 of course 1 and then on day 1 of all subsequent courses
  Standard analyses for the pharmacokinetic endpoints will be conducted, including summary of descriptive measures, e.g., tabulation of frequencies for categorical variables, numerical (mean, range, standard deviation, 95% confidence intervals) and graphical (box plots, histograms) summary of the distribution for continuous endpoints, correlation analyses (Pearson and Spearman), and linear and nonlinear regression analyses, etc.
Pharmacokinetic parameters of paclitaxel | On days 1, 2, 15, and 16 of course 1
  Standard analyses for the pharmacokinetic endpoints will be conducted, including summary of descriptive measures, e.g., tabulation of frequencies for categorical variables, numerical (mean, range, standard deviation, 95% confidence intervals) and graphical (box plots, histograms) summary of the distribution for continuous endpoints, correlation analyses (Pearson and Spearman), and linear and nonlinear regression analyses, etc.

OTHER OUTCOMES:
Change in expression of plasma markers | Baseline to up to day 17
  The marker expression will be compared by Student t-test.
PIK3CA mutation status | Up to day 17
  Chi-square or Fisher's exact status will be used to calculate associations between PIK3CA status and clinical parameters.
Prevalence of single nucleotide polymorphisms (SNPs) in PI3K pathway genes | Up to day 17
  Descriptive analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas